CLINICAL TRIAL: NCT03138213
Title: Total Laparoscopic Pancreaticoduodenectomy Versus Open Pancreaticoduodenectomy(TJDBPS01) a Multicenter Randomized Controlled Trial
Brief Title: Comparing Total Laparoscopic Versus Open Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government); The Second Hospital of Hebei Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Xinqiao Hospital of Chongqing (Other); Hunan Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The Third Affiliated Hospital of Soochow University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); First Affiliated Hospital of Chongqing Medical University (Other); Peking Union Medical College Hospital (Other); Henan Provincial People's Hospital (Other); Sir Run Run Shaw Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Clinical professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJDBPS01
Record Dates: First submitted 2017-02-07; First posted 2017-05-03 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Surgery; Periampullary Cancer
Keywords: pancreaticoduodenectomy; surgical outcome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLPD (Experimental): Ttotal laparoscopic pancreaticoduodenectomy
  Interventions: Procedure: Total laparoscopic pancreaticoduodenectomy
- OPD (Experimental): Open pancreaticoduodenectomy
  Interventions: Procedure: Open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Total laparoscopic pancreaticoduodenectomy — Total laparoscopic pancreaticoduodenectomy
  Arms: TLPD
Procedure: Open pancreaticoduodenectomy — Open pancreaticoduodenectomy
  Arms: OPD

SUMMARY:
Introduction Pancreatoduodenectomy (PD) is one of the most complex abdominal operations to perform, and it is usually conducted for tumours of the periampullary region and chronic pancreatitis. Minimally invasive surgery has been progressively being developed for pancreatic surgery, first with the advent of hybrid-laparoscopy and recently with total laparoscopic surgery. Issues including the safety and efficacy of total laparoscopic pancreaticoduodenectomy (TLPD) and open pancreaticoduodenectomy (OPD) are currently being debated. Studies comparing these two surgical techniques are emerging, and large randomized controlled trials (RCTs) are lacking but are clearly required.

Methods and analysis TJDBPS01 is a multicentre, prospective, randomized controlled, parallel-group, superiority trial in fourteen centres with pancreatic surgery experts who have performed ≥104 TLPDs and OPDs. A total of 656 patients who will undergo PD are randomly allocated to the TLPD group or OPD group in a 1:1 ratio. The trial hypothesis is that TLPD has superior or equivalent safety and advantages in postoperative recovery compared with OPD. The primary outcome is the postoperative length of stay (LOS).

Ethics and dissemination The Instituitional Review Board Approval of Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology has approved this trial and will be routinely monitoring the trial at frequent intervals, as will an independent third-party organization. Any results from this trial (publications, conference presentations) will be published in peer-reviewed journals and conference proceedings.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven periampullary cancer, including pancreatic cancer, bile duct cancer, duodenal cancer, et al.
2. Highly presumed malignancy with difficulties to obtain histological evidence.
3. Preoperative staging work up performed by upper abdomen enhanced CT scan.
4. The subject understands the nature of this trial and willing to comply.
5. Ability to provide written informed consent.
6. Patients treated with curative intent in accordance to international guidelines

Exclusion Criteria:

1. Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, involvement of other organs.
2. Subjects undergoing left, central or total pancreatectomy.
3. Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score >4.
4. Synchronous malignancy in other organs.
5. Previous underwent pancreatic resections.
6. Palliative surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | Up to 24 months
  Length of stay was defined as the postoperative time interval in days

SECONDARY OUTCOMES:
Estimated blood loss | Up to 24 months
  The amount of blood loss during surgical procedure.
Operation time | Up to 24 months
  Time between first incision and last skin closure.
Mortality | Up to 24 months
  Mortality was defined as any death that occurred in the 30 days after surgery or during the hospital stay.
Complication rate | Up to 24 months
  Clavien-Dindo
CCI | Up to 24 months
  comprehensive complication index
2 year survival | Up to 24 months
  Overall survival rate for 24 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin T, Zhang H, Pan S, Liu J, Li D, Chen R, Huang X, Liu Y, Liu J, Cheng W, Chen X, Zhao W, Li J, Tan Z, Huang H, Li D, Zhu F, Yu G, Zhou B, Zheng S, Tang Y, Ke J, Liu X, Chen B, Chen W, Ma H, Xu J, Liu Y, Lin R, Dong Y, Yu Y, Wang M, Qin R; Minimally Invasive Treatment Group in the Pancreatic Disease Branch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Effect of Laparoscopic and Open Pancreaticoduodenectomy for Pancreatic or Periampullary Tumors: Three-year Follow-up of a Randomized Clinical Trial. Ann Surg. 2024 Apr 1;279(4):605-612. doi: 10.1097/SLA.0000000000006149. Epub 2023 Nov 15. PMID 37965767
- [Derived] Wang M, Li D, Chen R, Huang X, Li J, Liu Y, Liu J, Cheng W, Chen X, Zhao W, Li J, Tan Z, Huang H, Li D, Zhu F, Qin T, Ma J, Yu G, Zhou B, Zheng S, Tang Y, Han W, Meng L, Ke J, Feng F, Chen B, Yin X, Chen W, Ma H, Xu J, Liu Y, Lin R, Dong Y, Yu Y, Liu J, Zhang H, Qin R; Minimally Invasive Treatment Group in the Pancreatic Disease Branch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Laparoscopic versus open pancreatoduodenectomy for pancreatic or periampullary tumours: a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Jun;6(6):438-447. doi: 10.1016/S2468-1253(21)00054-6. Epub 2021 Apr 27. PMID 33915091
- [Derived] Zhang H, Feng Y, Zhao J, Chen R, Chen X, Yin X, Cheng W, Li D, Li J, Huang X, Li J, Liu J, Liu J, Liu Y, Tan Z, Zhao W, Huang H, Li D, Yu Y, Wang M, Qin R. Total laparoscopic pancreaticoduodenectomy versus open pancreaticoduodenectomy (TJDBPS01): study protocol for a multicentre, randomised controlled clinical trial. BMJ Open. 2020 Feb 10;10(2):e033490. doi: 10.1136/bmjopen-2019-033490. PMID 32047015

DOCUMENTS (2):
  • Study Protocol (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03138213/Prot_003.pdf
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03138213/ICF_004.pdf